CLINICAL TRIAL: NCT06075537
Title: An Open-Label Extension to Investigate the Long-Term Safety, Tolerability, and Efficacy of DNL310 in Patients With Mucopolysaccharidosis Type II (MPS II) From Study DNLI-E-0002 or Study DNLI-E-0007
Brief Title: An Extension Study of the Long-Term Safety, Tolerability, and Efficacy of Tividenofusp Alfa (DNL310) in Participants With Mucopolysaccharidosis Type II (MPS II) From Study DNLI-E-0002 or Study DNLI-E-0007
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNLI-E-0008; 2023-503837-23 (Other: EU Trial Number)
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Mucopolysaccharidosis II
Keywords: Hunter Syndrome; MPS II; nMPS II; nnMPS II
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort A2 (Experimental): Participants with nMPS II, aged ≥5 to ≤10 years
  Interventions: Drug: tividenofusp alfa
- Cohort B2 (Experimental): Participants with nMPS II or nnMPS II, aged ≥1 to ≤18 years
  Interventions: Drug: tividenofusp alfa
- Cohort C2 (Experimental): Participants with nMPS II, aged <4 years
  Interventions: Drug: tividenofusp alfa
- Cohort D2 (Experimental): Participants with nMPS II or nnMPS II, aged ≤18 years with preexisting hepatomegaly who have never taken standard-of-care ERT
  Interventions: Drug: tividenofusp alfa
- Cohort E2 (Experimental): Participants with nMPS II, aged ≥6 years; participants with nnMPS II, aged <6 or ≥17 years; or participants with nMPS II, aged ≥1 to ≤18 years, with a history of prior HSCT or gene therapy and have completed at least 48 weeks in Study DNLI-E-0001
  Interventions: Drug: tividenofusp alfa
- Cohort A7 (Experimental): Participants with nMPS II, aged ≥2 to <6 years
  Interventions: Drug: tividenofusp alfa
- Cohort B7 (Experimental): Participants with nnMPS II, aged ≥6 to <17 years
  Interventions: Drug: tividenofusp alfa

INTERVENTIONS:
Drug: tividenofusp alfa — Intravenous repeating dose

SUMMARY:
This is a multiregional open-label extension (OLE) to assess the safety, tolerability, and efficacy of long-term treatment with tividenofusp alfa (DNL310), an investigational central nervous system (CNS)-penetrant intravenous (IV) enzyme replacement therapy (ERT) for Hunter syndrome (MPS II). Participants who complete at least through the Week 49 visit in Study DNLI-E-0002 and do not discontinue study intervention early and participants who complete Study DNLI-E-0007 will be enrolled in this OLE. All participants will receive DNL310 for up to 5 years from the time of entry in this OLE. Participants, site staff, and the Sponsor will remain blinded to the original treatment assignment for participants entering this OLE from Study DNLI-E-0007.

ELIGIBILITY:
Key Inclusion Criteria:

* For participants from Study DNLI-E-0002 only: Completed at least through the Week 49 visit in Study DNLI-E-0002 and did not discontinue study intervention early
* For participants from Study DNLI-E-0007 only: Completed the treatment period of 96 weeks in Cohort A for nMPS II participants and 48 weeks in Cohort B for nnMPS II participants

Key Exclusion Criteria:

* Unstable or poorly controlled medical condition(s) or significant medical or psychological comorbidity or comorbidities that, in the opinion of the investigator, would interfere with safe participation in the trial or interpretation of study assessments

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and intensity of treatment-emergent adverse events (TEAEs) | 5 years
Clinically significant changes in urine total glycosaminoglycan (GAG) concentrations throughout the treatment period | 5 years
Incidence and intensity of infusion-related reactions (IRRs) | 5 years
  The intensity of IRRs will be assessed following each infusion of DNL310 using the categories of Mild, Moderate and Severe. IRRs will be summarized overall as well as stratified by intensity.

SECONDARY OUTCOMES:
Percentage change from baseline in cerebrospinal fluid (CSF) heparan sulfate (HS) concentration | 5 years
Change from baseline in the Vineland-3 Adaptive Behavior Scale | 5 years
Change from baseline in the Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) cognitive raw score | 5 years
Change from baseline in distance walked (meters) in the Six-Minute Walk Test (6MWT) | 5 years
Percent change from baseline in the sum of urine HS and dermatan sulfate (DS) concentrations | 5 years
Liver volume within the normal range (normal vs abnormal) as measured by MRI | 5 years
Spleen volume within the normal range (normal vs abnormal) as measured by MRI | 5 years
Improvement in the Parent/Caregiver Global Impression of Change (CaGI-C) Overall MPS II | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose Alcantara Rodriguez, PharmD, Study Director — Denali Therapeutics
Locations (22):
- United States (6):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UNC Children's Research Institute, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Medical School at Houston, Houston, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
- Sanatorio Mater Dei, Buenos Aires, Argentina
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - UZ Brussel, Jette
- Canada (3):
  - University of Alberta - Faculty of Medicine & Dentistry, Edmonton, Alberta
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- Vseobecna Fakultni Nemocnice V Praze, Prague, Czechia
- Hopital Jeanne De Flandre - Metabolic Diseases Unit, Lille, France
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - SpinCS GmbH, Höchheim
- Azienda Sanitaria Universitaria Friuli Centrale - PO Universitario Santa Maria della Misericordia, Udine, Italy
- Erasmus Medical Center - Sophia Children's Hospital, Rotterdam, Netherlands
- Hospit U. Vall d'Hebron - PPDS, Barcelona, Spain
- Drottning Silvias Barn Och Ungdomssjukhus, Gothenburg, Sweden
- Turkey (Türkiye) (2):
  - University Medical Faculty Balcali Hospital, Adana
  - Gazi Universitesi Tip Fakultes, Ankara

IPD SHARING:
Plan to Share IPD: No